CLINICAL TRIAL: NCT03579108
Title: Hypertension Management and Outcomes in a Family Practice Setting
Brief Title: Hypertension Management in Family Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Erwin A. Aguilar, Associate Professor, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: LSUIRB 9976
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective Chart Review — Chart review
  Other Names: Chart review

SUMMARY:
High blood pressure is the greatest threat to the global burden of disease, contributing to an estimated 9.4 million deaths a year. Cardiovascular disease morbidity and mortality are positively correlated with the degree of elevation of blood pressure, without any evidence of a threshold down to at least 115/75 mm Hg[2]. Hypertension is common, and nearly every clinician in every specialty deals either directly or indirectly with managing it or its consequences.

The population age 65 years or older numbered 46.2 million in 2014 and they represent 14.5% of the US population, the older population in 2030 is projected to be more than twice as large as in 2000, growing from 35 million to 74 million and representing 21 percent of the total U.S. population and it is expected to more than double to 98 million in 2060.Proper managing and controlling blood pressure markedly improves patient morbidity and mortality, SHEP study showed that in persons aged 60 years and over with isolated systolic hypertension, antihypertensive stepped-care drug treatment with low-dose chlorthalidone as step 1 medication reduced the incidence of total stroke by 36%.This study will estimate the prevalence of hypertension diagnosis, treatment and outcomes in a Family Practice population. It is a hypothesis generating study

DETAILED DESCRIPTION:
This a retrospective cross-sectional chart review study. The study population will consist of a random sample of patients from the Family Practice of the LSU Department of Family Medicine at LSU Health Sciences Center in New Orleans (LSUHSC-NO) Chart data will be collected retrospectively back to one year from date of starting data abstraction.

Data Quality The data used in this study comes from patient charts that are actively being used in the management of patient care. Data quality will be ensured through several means. First, the data collection process will be conducted family medicine resident. Second, data will be abstracted directly into an electronic encrypted Excel file.

Selection of Participants The family medicine residents will take each one 25 patients each and review the charts and record the information on an Excel spread sheet.

ELIGIBILITY:
Inclusion Criteria

* hypertension

Exclusion Criteria:

* No hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family Medicine Practice
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-24 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
controlled hypertension | 3 months
  number of patients controlled and non controlled

CONTACTS AND LOCATIONS:
Overall Officials: Erwin A Aguilar, PharmD, MPH, Principal Investigator — LSU Health Sciences Center in New Orleans
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Statistics, F. I.-R. (2016). Older Americans 2016: Key Indicators of Well-Being. Washington, DC: Federal Interagency Forum on Aging-Related Statistics. Retrieved from AgingStats.gov
- [Background] HHS. (2015). A profile of Older Americans: 2015. Washingtin, D.C: HHS. Retrieved from Profile of Older American.
- [Background] Ostchega Y, Dillon CF, Hughes JP, Carroll M, Yoon S. Trends in hypertension prevalence, awareness, treatment, and control in older U.S. adults: data from the National Health and Nutrition Examination Survey 1988 to 2004. J Am Geriatr Soc. 2007 Jul;55(7):1056-65. doi: 10.1111/j.1532-5415.2007.01215.x. PMID 17608879
- [Background] Butt DA, Harvey PJ. Benefits and risks of antihypertensive medications in the elderly. J Intern Med. 2015 Dec;278(6):599-626. doi: 10.1111/joim.12446. Epub 2015 Oct 26. PMID 26497967
- [Background] Franklin SS, Jacobs MJ, Wong ND, L'Italien GJ, Lapuerta P. Predominance of isolated systolic hypertension among middle-aged and elderly US hypertensives: analysis based on National Health and Nutrition Examination Survey (NHANES) III. Hypertension. 2001 Mar;37(3):869-74. doi: 10.1161/01.hyp.37.3.869. PMID 11244010
- [Background] Buford TW. Hypertension and aging. Ageing Res Rev. 2016 Mar;26:96-111. doi: 10.1016/j.arr.2016.01.007. Epub 2016 Feb 1. PMID 26835847
- [Background] Franklin SS, Gustin W 4th, Wong ND, Larson MG, Weber MA, Kannel WB, Levy D. Hemodynamic patterns of age-related changes in blood pressure. The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):308-15. doi: 10.1161/01.cir.96.1.308. PMID 9236450
- [Background] Kjeldsen S, Feldman RD, Lisheng L, Mourad JJ, Chiang CE, Zhang W, Wu Z, Li W, Williams B. Updated national and international hypertension guidelines: a review of current recommendations. Drugs. 2014 Nov;74(17):2033-51. doi: 10.1007/s40265-014-0306-5. PMID 25315030
- [Background] Go AS, Bauman MA, Coleman King SM, Fonarow GC, Lawrence W, Williams KA, Sanchez E; American Heart Association; American College of Cardiology; Centers for Disease Control and Prevention. An effective approach to high blood pressure control: a science advisory from the American Heart Association, the American College of Cardiology, and the Centers for Disease Control and Prevention. Hypertension. 2014 Apr;63(4):878-85. doi: 10.1161/HYP.0000000000000003. Epub 2013 Nov 15. No abstract available. PMID 24243703
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Reisin E, Harris RC, Rahman M. Commentary on the 2014 BP guidelines from the panel appointed to the Eighth Joint National Committee (JNC 8). J Am Soc Nephrol. 2014 Nov;25(11):2419-24. doi: 10.1681/ASN.2014040371. Epub 2014 Aug 11. PMID 25114277
- [Background] Weber MA, Schiffrin EL, White WB, Mann S, Lindholm LH, Kenerson JG, Flack JM, Carter BL, Materson BJ, Ram CV, Cohen DL, Cadet JC, Jean-Charles RR, Taler S, Kountz D, Townsend R, Chalmers J, Ramirez AJ, Bakris GL, Wang J, Schutte AE, Bisognano JD, Touyz RM, Sica D, Harrap SB. Clinical practice guidelines for the management of hypertension in the community a statement by the American Society of Hypertension and the International Society of Hypertension. J Hypertens. 2014 Jan;32(1):3-15. doi: 10.1097/HJH.0000000000000065. No abstract available. PMID 24270181
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Dasgupta K, Quinn RR, Zarnke KB, Rabi DM, Ravani P, Daskalopoulou SS, Rabkin SW, Trudeau L, Feldman RD, Cloutier L, Prebtani A, Herman RJ, Bacon SL, Gilbert RE, Ruzicka M, McKay DW, Campbell TS, Grover S, Honos G, Schiffrin EL, Bolli P, Wilson TW, Lindsay P, Hill MD, Coutts SB, Gubitz G, Gelfer M, Vallee M, Prasad GV, Lebel M, McLean D, Arnold JM, Moe GW, Howlett JG, Boulanger JM, Larochelle P, Leiter LA, Jones C, Ogilvie RI, Woo V, Kaczorowski J, Burns KD, Petrella RJ, Hiremath S, Milot A, Stone JA, Drouin D, Lavoie KL, Lamarre-Cliche M, Tremblay G, Hamet P, Fodor G, Carruthers SG, Pylypchuk GB, Burgess E, Lewanczuk R, Dresser GK, Penner SB, Hegele RA, McFarlane PA, Khara M, Pipe A, Oh P, Selby P, Sharma M, Reid DJ, Tobe SW, Padwal RS, Poirier L; Canadian Hypertension Education Program. The 2014 Canadian Hypertension Education Program recommendations for blood pressure measurement, diagnosis, assessment of risk, prevention, and treatment of hypertension. Can J Cardiol. 2014 May;30(5):485-501. doi: 10.1016/j.cjca.2014.02.002. Epub 2014 Feb 22. PMID 24786438
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F, Redon J, Dominiczak A, Narkiewicz K, Nilsson PM, Burnier M, Viigimaa M, Ambrosioni E, Caufield M, Coca A, Olsen MH, Schmieder RE, Tsioufis C, van de Borne P, Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S, Clement DL, Coca A, Gillebert TC, Tendera M, Rosei EA, Ambrosioni E, Anker SD, Bauersachs J, Hitij JB, Caulfield M, De Buyzere M, De Geest S, Derumeaux GA, Erdine S, Farsang C, Funck-Brentano C, Gerc V, Germano G, Gielen S, Haller H, Hoes AW, Jordan J, Kahan T, Komajda M, Lovic D, Mahrholdt H, Olsen MH, Ostergren J, Parati G, Perk J, Polonia J, Popescu BA, Reiner Z, Ryden L, Sirenko Y, Stanton A, Struijker-Boudier H, Tsioufis C, van de Borne P, Vlachopoulos C, Volpe M, Wood DA. 2013 ESH/ESC guidelines for the management of arterial hypertension: the Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Eur Heart J. 2013 Jul;34(28):2159-219. doi: 10.1093/eurheartj/eht151. Epub 2013 Jun 14. No abstract available. PMID 23771844
- [Background] Jaques H; National Institute for Health and Clinical Excellence (NICE). NICE guideline on hypertension. Eur Heart J. 2013 Feb;34(6):406-8. No abstract available. PMID 23520636
- [Background] American Diabetes Association. (8) Cardiovascular disease and risk management. Diabetes Care. 2015 Jan;38 Suppl:S49-57. doi: 10.2337/dc15-S011. No abstract available. PMID 25537708
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Prevention of stroke by antihypertensive drug treatment in older persons with isolated systolic hypertension. Final results of the Systolic Hypertension in the Elderly Program (SHEP). SHEP Cooperative Research Group. JAMA. 1991 Jun 26;265(24):3255-64. PMID 2046107